CLINICAL TRIAL: NCT04637256
Title: Evaluation of Outcomes from Treatment of Benign or Malignant Gastroesophageal Diseases
Status: Recruiting | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 037.HPB.2018.R
Record Dates: First submitted 2019-03-22; First posted 2020-11-19 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-08

CONDITIONS: Pancreatic Malignant Neoplasm Primary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study will be a retrospective chart review of patients who have been diagnosed with benign or malignant pancreatic disease under the practice of Dr. Rohan Jeyarajah, M.D., Dr. Houssam Osman M.D., and Dr. Edward Cho M.D., Sc.M. at Methodist Health System Hospital in Richardson, TX. The Investigators plan to conduct an analysis of patients meeting the inclusion criteria from 2005 to present. Study will also be conducted by the PI, Sub-Is, surgery fellows, office staff and clinical research coordinator who are delegated to do by the PI. Data will be obtained by looking through either the investigator's patients from their practice or through a national database. Data will be analyzed primarily by the study conductors.

DETAILED DESCRIPTION:
1. INTRODUCTION 1.1. Background It is reported in the literature that the treatment of any gastroesophageal disease process, whether benign or malignant, continues to be a huge challenge. For example, patients with esophageal cancer continue to be diagnosed at an advanced stage with medical and surgical options that are improving in terms of outcome measurements but with much more room for improvement. The Primary investigtor goal is to continue to review patient treatment outcomes to further improve overall survival, overall symptom control, mortality and morbidity.

1.2. Aim(s)/Objective(s) The main aim of this study is to evaluate and compare the outcomes from the investigator's treatment of benign or gastroesophageal diseases.

1.3. Rationale for the study There is a need to understand and improve the current diagnosis and treatment algorithm for gastroesophageal pathologies. Continued evaluation and study is imperative to ensure that national guidelines are improving to enhance patient cure and/or recovery.

2. OBJECTIVES AND STUDY OUTCOME MEASURES 2.1. Study Objectives 2.1.1. Primary Objective(s)

• To evaluate and compare the outcomes from the investigator's treatment of benign or malignant gastroesophageal disease 2.2. Study Outcome Measures 2.2.1. Primary Outcome(s)

* To exam all treatments of benign or malignant gastroesophageal disease by measuring the following outcomes o Overall survival o Overall symptom control

  o Mortality

  o Morbidity 4. STUDY ENROLLMENT AND WITHDRAWAL 4.1. Study Inclusion Criteria:
* All patients diagnosed and treated for gastroesophageal diseases, benign or malignant from 2005 to present.
* Age ≥18 years 4.2. Study Exclusion Criteria:
* Patients that are not diagnosed with or treated for gastroesophageal diseases
* Age < 18 years 5. STATISTICAL CONSIDERATIONS 5.1. Sample Size Considerations All past patients who were treated for a particular benign or malignant gastroesophageal disease process under evaluation from 2005 to present will be included in this study.

5.2. Statistical Analysis Plan Statistics will be provided for all data obtained. Normally distributed continuous outcomes will be analyzed with Student's t test and non-normally distributed continuous outcomes will be analyzed with nonparametric Wilcoxon-Mann-Whitney test. Categorical outcomes will be analyzed using chi-square test or Fisher's exact test for smaller samples.

6. ETHICS/PROTECTION OF HUMAN SUBJECTS 6.1. Ethical Standard 6.1.1. The following safeguard will be employed to protect confidentiality of data

* Limitation of access to data
* Minimal HIPAA identifiers on data collection tools
* Password protected share drive database on computer
* Use of locked file cabinets for physical records (if any collected)
* Restricted access to share drive database on computers
* Appropriate training of personnel accessing share drive database
* At close of this study, all identifiers will be removed from the data collection tools 6.2. Institutional Review Board The protocol and all study related materials will be submitted to the IRB for review and approval. Approval of both the protocol and study related material will be obtained before any clinical data is collected. Any amendment to the protocol will require review and approval by the IRB before the changes are implemented in the study.

6.3. Informed Consent Process 6.3.1. Details to waive consent for this retrospective chart review

• This research is not regulated by the FDA

* The research involves no more than minimal risk to the subjects
* The waiver or alternation will not adversely affect the rights or welfare of the subjects
* The research could not practicably be carried out without the waiver
* It is not feasible to provide subjects with pertinent information after participation 6.4. Participant Confidentiality
* All data collection will be kept in password protected hospital server
* Only authorized personal will have access share drive
* Patient confidentiality will be maintained at all times, complying with HIPAA guidelines.

  7. DATA MANAGEMENT PLAN 7.1. Source Document Management

The investigator(s)/institution(s) will permit study-related monitoring, audits, IEC/IRB review, and regulatory inspection(s), providing direct access to data collected via the Methodist Health System share drive. Data collected during this study will be recorded on the appropriate data source via word document, access database, and excel spread sheet depending on treatment type capturing the following data but not limited to:

* • Demographics

  * Subject number
  * First and Last Name
  * Medical Record Number
  * Social Security
  * Gender
  * Ethnicity
  * Race
  * Date of Birth
* Diagnosis

  * Date of Diagnosis
  * Age at Diagnosis
  * Class of Case
  * Symptoms Associated with Diagnosis Onset date Length of Symptom On set
  * Eckcardt Score
  * Clinical T
  * Clinical N
  * Clinical M
  * Clinical Stage
  * R Status
  * Pre-Op Work Up and Results
  * Date of 1st Contact
  * Zip code at Diagnosis
* Medical History

  * Diagnosis
  * On set Date
* Medication List

  * Name
  * Dose
  * Frequency
* Social Medical History

  * Depression
  * Tobacco Never Smoked Current Smoker
* Amount of Cigarettes per day/week Ex-Smoker
* Date of Quitting
* Amount of Cigarettes per day/week

  o Alcohol Never Consumed Alcohol
* Amount of consumption per day/week/month Current Alcohol User
* Amount of consumption per day/week/month

  * Jaundice
  * Drug/ Substance Abuse
  * Reported Weight Loss Weight lbs. and kg. Length of Weight Loss on set
* Anesthesia

  * Type of Anesthesia
  * ASA
  * Anesthesia Start and End Time
  * Medication list Name Dose Frequency
  * Intra-Ops I/O's
  * Est. Blood loss (ml)
  * Blood Transfusions
  * Patient Position
  * Complication
  * Notes
* Surgery

  * Date
  * Age at Surgery Visit
  * Pre-op Stent
  * TPN
  * Primary Site
  * Classification of Diagnosis
  * Pre-Op Diagnosis
  * Post-Op Diagnosis
  * Proposed Procedure
  * Actual Procedure
  * Laparoscopic
  * Laparotomy
  * Pylorus preserved
  * Procedure Start and end time
  * Operative time
  * Prophylactic antibiotic
  * Intra-op antibiotic redoes
  * Ng tube
  * Adjusted Est. Blood Loss
  * Est. Blood loss (ml)
  * Drains inserted
  * Specimens Collected
  * Specimen Results
  * Complications
  * Hospital and Discharge Medication List
  * Name
  * Dose
  * Frequency
  * Post Medication List
  * Name
  * Dose
  * Frequency
* Vitals

  o In the following times points: Pre-Op, Intra-Op, Post-Op, and Discharge Systolic Diastolic Pulse rate Temperature Respiration BMI
* Lab

  * In the following time points: Pre-op and Post-op at different F/U Visit AST ALT ALP TOTAL BILIRUBIN DIRECT BILIRUBIN TOTAL PROTEIN PRE ALBUMIN ALBUMIN CA 19-9 CEA CRP WBC/ LEUKOCYTES HGB HCT MCV PLATELETS BIOCARBONATE (TOTAL CO2) AFP AMYLASE LIPASE JP AMYLASE
* Pathology

  * Final Diagnosis
  * Diagnosis Comment
  * Clinical Information
  * Gross Description
  * Microscopic Description
  * Diagnosis histology
  * Benign/malignant
  * Pathology T
  * Pathology N
  * Pathology M
  * Pathology Stage
  * R status
  * Grade
  * Tumor size (cm)
  * All Margins
  * All Lymph Nodes
  * Perineural invasion
  * Lymph invasion
  * Vascular invasion
  * SPN LN
  * LBD LN
  * Regional LN examined
  * Regional LN positive
* Imaging

  * Pre-op CT Date of Exam Type of Exam Findings/Impressions
  * Pre-op MRI Date of Exam Type of Exam Findings/Impressions
  * Pre-op PET Date of Exam Type of Exam Findings/Impressions
  * Post-op CT at Different F/U Visit Date of Exam Type of Exam Findings/Impressions
  * Post-op MRI at Different F/U Visit Date of Exam Type of Exam Findings/Impressions
  * Post-op PET at Different F/U Visit Date of Exam Type of Exam Findings/Impressions
* Inpatient

  * Admission date
  * Discharge date
  * LOS (days)
  * LOS after surgery (days)
  * Direct floor transfer
  * ICU stay
  * ICU admission date
  * ICU discharge date
  * Length of ICU stay (days)
  * Tube feed
  * TF #
  * TF start date
  * TF end date
  * TF Post-OP
  * Oral
  * Oral start date
  * Oral post-op
  * Reglan
  * Entereg
  * Entereg 1st oral intake
  * Bowel movement date
  * Time to 1st of bowel movement (days)
  * Medication list Name Dose Frequency
  * Complications
  * Discharge Diagnosis
* Complications

  * Readmit within 30 days of d/c
  * Reason for readmit
  * Delayed gastric emptying
  * Pancreatic fistula
  * Wound infection
  * Intraabdominal abscess
  * Cardiac event
  * Pancreatitis
  * Bile leak
  * Pneumonia
  * Hemobilia
  * Lymphatic leak
  * Pancreatic leak
  * GI bleed
  * Anemia
  * Reoperation
  * Other morbidities
* Comorbidities

  * Cerebrovascular Accident
  * Peripheral Vascular Disease
  * Diabetes
  * Hypertension
  * MYO Card Infarct
  * COPD
  * Malnutrition
  * CHF
  * Revised co-morb scale
  * Other
* Pre-Op and Post-op Chemo and Radiation o Chemo start date

  o Chemo end date
  * Chemo regimen
  * # of completed cycles
  * Pre-op or post-op or both
  * Patient declined
  * Contraindicated
  * Course date radiation started
  * Course date radiation ended
  * Dose
  * Fractions
* Post Op Follow up Clinical/Phone Visit

  o Follow Up Visit Date
  * Symptoms Reported
  * Length of Symptom On set
  * Medication list Name Dose Frequency
  * Eckcardt Score
* Patient Outcome o Site of recurrence

  o Date of recurrence

  o Clinical/path dx recurrence

  o Recurrence
  * Recurrence Surgery Date
  * Disease free
  * Follow up
  * Date of death
  * Post op mortality

7.2. Data Capture Methods • Data will be collected and entered at MRMC

• Data will be captured from Methodist Health System eMAR and TSC Clinical eMAR

• A secure Methodist Health System share drive will host all data

• Training and access to share drive will be given to all study staff as delegated per PI

• Data collected during this study will be recorded on the appropriate data source via word document, access database, and/or excel spread sheet depending on treatment type capturing the following data but not limited to demographics, treatment, pre-operative evaluation, surgical technique, hospitalization, and post-operative evaluation. Stored insecure share drive with access limited to study staff in a password protected computer at MRMC

8. PUBLICATION PLAN All information will be blinded in compliance with GCP. The investigator will make all possible efforts to ensure compliance with all policies regarding sharing of PHI or research information. Only de-identified PHI will be shared in relevant research mediums. These mediums may range from national, regional, local and/or international sites. In addition, study data and findings may be submitted for presentation at local and national conferences

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed and treated for gastroesophageal diseases, benign or malignant from 2005 to present.
* Age ≥18 years

Exclusion Criteria:

* Patients that are not diagnosed with or treated for gastroesophageal diseases
* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All past patients who were treated for a particular benign or malignant gastroesophageal disease process under evaluation from 2005 to present will be included in this study.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-03-06 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 2005 to 2019
  We will be examining all treatments of benign or malignant pancreatic cancer by measuring the following outcome: overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Dhiresh Jeyarajah, M.D., Principal Investigator — Methodist Health System
Locations (1):
- Trinity Surgical Consultants, Methodist Richardson Medical Center, Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: No